CLINICAL TRIAL: NCT05744895
Title: Early Outcomes of Total Knee Arthroplasty Using the MAKO Surgical Robot and Triathlon Knee
Brief Title: MAKO Total Knee Artroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: 202106145
Record Dates: First submitted 2023-02-01; First posted 2023-02-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Prospective Group- Robotic TKA Arm: Prospective TKA patient receiving total knee arthroplasty using the MAKO robotic machine
  Interventions: Device: Device: Robotic MAKO total knee; Device: FocusMotion knee brace; Device: Fitbit tracking device; Device: FocusMotion app
- Control- manual total Knee arthroplasty: Patients who have had a manual total knee arthroplasty

INTERVENTIONS:
Device: Device: Robotic MAKO total knee — Prospective TKA patient receiving total knee arthroplasty using the MAKO robotic machine
  Groups: Prospective Group- Robotic TKA Arm
Device: FocusMotion knee brace — Focusmotion knee brace measures range of motion during exercises
  Groups: Prospective Group- Robotic TKA Arm
Device: Fitbit tracking device — Fitbit will measure patients steps, HR, and sleep
  Groups: Prospective Group- Robotic TKA Arm
Device: FocusMotion app — Will survey patients with PROMS
  Groups: Prospective Group- Robotic TKA Arm

SUMMARY:
The purpose of this study is to determine the early clinical and radiographic outcomes of robotically assisted total knee arthroplasty with the MAKO surgical robot using the Triathlon knee system. Results of this study will be compared to those of a previously published cohort of patients from this institution who underwent TKA using non-robotic, manual instruments.

MAKO TKA patients will be given Fitbits and the Focus Motion Knee Brace to capture the data listed in attachment section. The results of this data will be compared to the control group to see if there is or there is not a difference in clinical outcomes with patients receiving Total knee surgery using the MAKO surgical robot versus those who got Total knee surgery without the MAKO robot.

DETAILED DESCRIPTION:
Research objectives:

The purpose of this study is to determine the early clinical and radiographic outcomes of robotically assisted total knee arthroplasty with the MAKO surgical robot using the Triathlon knee system. Mean weekly VAS pain score during the first 4 weeks is the primary end point. Results of this study will be compared to prospective cohort of patients in the IRB study 201805014 from this institution who underwent TKA using non-robotic, manual instruments

Primary Hypothesis: Patients receiving robotic TKA will have better early recovery, including lower mean weekly VAS pain score for the first 4 weeks postoperatively and higher functional outcome scores, than the manual TKA historical cohort.

Secondary Hypothesis:

Patients receiving robotic TKA will have more accurate component position and alignment than the manual TKA historical cohort.

Potential Contribution: This study would give us a better understanding of the clinical and radiographic outcomes of patients receiving robotic TKA versus manual TKA. It will identify potential advantages and disadvantages of robotic TKA using the MAKO surgical robot.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo Unilateral primary total knee arthroplasty
* 18 and up
* Willing to sign informed consent
* Willing to return for all follow-up visits
* Smartphone or tablet device capable of running the Fitbit andFocusMotion platform

Exclusion Criteria:

* BMI > 45
* Inflammatory arthritis
* Narcotic use greater than 5 days per week
* Walking aid for musculoskeletal or neurologic issue other than operative joint
* Bilateral total knee arthroplasty
* Patient with an active infection or suspected infection in the operative joint
* The absolute and relative contraindications stated in the FDA cleared labeling for the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We propose to enroll patients that are scheduled for a MAKO Total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Early recovery | 4 weeks
  To determine if Robotic-arm assisted TKA (RA-TKA) allows for earlier recovery than manual TKA (MI-TKA). This will be measured by weekly VAS pain score.
  [Time Frame: 1 day- post op]

SECONDARY OUTCOMES:
Post op EOS measurements for alignment | 1 year
  To determine if Robotic-arm assisted TKA (RA-TKA) allows for more accurate component placement than manual TKA (MI-TKA). units of measurement will be inches.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hannon, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Creve Coeur, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT05744895/Prot_000.pdf